CLINICAL TRIAL: NCT02095691
Title: A Prospective, Multi-center, Non-Randomized, Feasibility Study of Catheter Based Renal Denervation to Treat Resistant Hypertension (RENABLATE-II - 157)
Brief Title: RENABLATE-II Feasibility Study of Catheter Based Renal Denervation to Treat Resistant Hypertension - 157
Acronym: RENABLATE-II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENABLATE-II
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Renal
Keywords: Renal Sympathetic Denervation
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistant Hypertension (Experimental): The Celsius® ThermoCool® Renal Denervation catheter will serve to treat resistant hypertension.
  Interventions: Device: Celsius® ThermoCool® Renal Denervation

INTERVENTIONS:
Device: Celsius® ThermoCool® Renal Denervation — The investigational device is indicated for the treatment of resistant hypertension by renal denervation.
  Other Names: Multi-electrode Ablation Catheter

SUMMARY:
This is a prospective, multi-center, non-randomized, feasibility study to assess the safety and effectiveness of renal artery sympathetic denervation using the investigational devices in subjects with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a systolic blood pressure ≥ 140 mmHg based on an average of 3 office blood pressure readings measured according to the BP guidelines.
2. Subject is adhering to a stable drug regimen of at least 3 different classes of anti-hypertensive medications, including a diuretic (with no changes for a minimum of 2 weeks prior to enrollment) at optimal dose and is expected to be maintained for at least 6 months.
3. Subject is > 18 and < 85 years of age.
4. Subject agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this study.

Key Exclusion Criteria:

1. A secondary cause of hypertension, e.g. "white coat" hypertension (assessed by 24 h ABPM at physician's discretion), primary aldosteronism, pheochromocytoma, renal artery stenosis, drug induced-hypertension, Adult Polycystic kidney Disease, renal cell carcinoma, pyelonephritis, glomerulonephritis, coarctation of the aorta, acromegaly, Cushing's Syndrome, Conn's (primary hyperaldosteronism), polyarteritis nodosum, systemic sclerosis, parenchymal kidney disease, obstructive sleep apnoea based on a workup performed within the 12 months preceding enrollment.
2. Subject has aorto-ilio-femoral artery anatomy not suitable for treatment with the investigational device(s).
3. Subject has main renal arteries that are < 20 mm in length or < 4 mm in diameter.
4. Subject has a prior history of any renal artery intervention including but not limited to balloon angioplasty, stenting, renal denervation or surgery.
5. Subject has an estimated glomerular filtration rate (eGFR) of < 45mL/min/1.73m2, using the MDRD formula.
6. Subject has type 1 diabetes mellitus.
7. Subject has history of Myocardial Infarction, unstable angina pectoris, or a cerebrovascular accident in the 6 months period prior to enrolment, or documented widespread atherosclerosis, intravascular thrombosis or unstable plaques.
8. Subject has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2015-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrollment took approximately 3 months, began on October 21, 2013 and completed on December 17, 2013. A total of 37 subjects were consented and 19 underwent treatment with the study catheter in 4 investigation sites in New Zealand, Czech Republic, and Italy.
Groups:
- Renal Artery Sympathetic Denervation: Subjects enrolled in this study underwent the renal artery sympathetic denervation procedure for treating moderate resistant hypertension. The procedure was conducted with the investigational Celsius® ThermoCool® Renal Denervation catheter.
Period: Overall Study
Arm/Group | Renal Artery Sympathetic Denervation
Started | 19 (Subjects who were consented and treated with study ablation catheter.)
Completed | 18 (Subjects with follow up available at 12 months.)
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis population which consists of all enrolled subjects who have undergone insertion of the study ablation catheter.
Arm/Group | Renal Artery Sympathetic Denervation
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  African Descent | 1
  Not African Descent | 18
Region of Enrollment [Number; unit: participants]
  New Zealand | 6
  Czech Republic | 9
  Italy | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Major Adverse Events That Occurred Within 30 Days Post-procedure.
Description: Major adverse events include Acute myocardial infarction; Death from progressive heart failure, death from aortic or peripheral artery disease, from renal failure and sudden cardiac death; New-onset heart failure; Stroke; Aortic or lower limb revascularization procedure; Lower limb amputation; Beginning dialysis; Hospital admission for hypertensive emergency unrelated to non-adherence or non-persistence with drugs at each follow up visit; Hospitalization for atrial fibrillation.
Time Frame: 30 days post-procedure
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Renal Artery Sympathetic Denervation
Number analyzed (Participants) | 19
percentage of participants | 0.0

2. Secondary Outcome: Incidence of Adverse Cardiovascular and Renal Events Within the 12 Month Follow-up Visit
Description: These adverse events include renal artery stenosis (≥60% diameter reduction confirmed by MRI or renal angiography); peri-procedural renal artery dissection or perforation requiring intervention, serious arterial access site related complications requiring intervention or prolonging hospitalization; ≥25% reduction between baseline and 12 months in renal function measured by the estimated Glomerular Filtration Rate (eGFR), as well as composite of major adverse cardiovascular and/or renal events.
Time Frame: 12 months post-procedure
Population: The safety analysis population consists of all enrolled subjects who have undergone insertion of the study ablation catheter.
Measure: Number; unit: percentage of participants
Arm/Group | Renal Artery Sympathetic Denervation
Number analyzed (Participants) | 19
percentage of participants | 42.1

3. Secondary Outcome: Mean Change in Office Systolic Blood Pressure and Diastolic Blood Pressure From Baseline to 1 ,3, 6 and 12 Months Post Procedure
Description: Office systolic blood pressure (SBP) and diastolic blood pressure (DBP) measures were summarized to assess the reduction in blood pressure from baseline visit to post baseline at 1, 3, 6, and 12 months. Negative values for change represent reductions.
Time Frame: 12 months post-procedure
Population: Effectiveness analysis population, which consists of enrolled subjects without enrollment deviation and experiencing technical success. Technical success is defined as the investigational catheter being successfully inserted into the femoral artery with radiofrequency energy successfully applied in at least one artery.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Change in Blood Pressure at 1 Month Follow up: Change in Blood Pressure from baseline to1 month follow up
- Change in Blood Pressure at 3 Months Follow Up: Change in Blood Pressure from baseline to3 months follow up
- Change in Blood Pressure at 6 Months Follow Up: Change in Blood Pressure from baseline to 6 months follow up
- Change in Blood Pressure at 12 Month Follow Up: Change in Blood Pressure from baseline to 12 months follow up
Arm/Group | Change in Blood Pressure at 1 Month Follow up | Change in Blood Pressure at 3 Months Follow Up | Change in Blood Pressure at 6 Months Follow Up | Change in Blood Pressure at 12 Month Follow Up
Number analyzed (Participants) | 14 | 14 | 14 | 13
mmHg
  Mean Reduction in SBP | -16.4 (18.3) | -14.5 (25.1) | -11.3 (24.4) | -13.8 (23.9)
  Mean Reduction in DBP | -10.1 (12.1) | -5.2 (11.7) | -1.3 (10.2) | -4.9 (10.3)

4. Secondary Outcome: Incidence of Subjects Achieving Target Systolic Blood Pressure (SBP) at 1, 3, 6 and 12 Months Post Procedure
Description: The pre-specified target SBP is defined as SBP <130 mmHg. This endpoint is defined at each of 1, 3, 6 and 12 months post procedure.
Time Frame: 12 months post-procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- At 1 Month Follow up: Percentage of subjects achieving target SBP at 1 month follow up
- At 3 Months Follow Up: Percentage of subjects achieving target SBP at 3 months follow up
- At 6 Months Follow Up: Percentage of subjects achieving target SBP at 6 months follow up
- At 12 Month Follow Up: Percentage of subjects achieving target SBP at 12 months follow up
Arm/Group | At 1 Month Follow up | At 3 Months Follow Up | At 6 Months Follow Up | At 12 Month Follow Up
Number analyzed (Participants) | 14 | 14 | 14 | 13
percentage of participants | 28.6 | 7.1 | 7.1 | 7.1

5. Secondary Outcome: Incidence of Subjects Achieving a ≥ 10 mmHg Reduction in Systolic Blood Pressure (SBP) at 1, 3, 6 and 12 Months Post Procedure
Description: Incidence of subjects achieving a 10 mmHg or more reduction in Systolic Blood Pressure (SBP) at 1, 3, 6 and 12 months post procedure.
Time Frame: 12 months post-procedure
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- At 1 Month Follow up: Percentage of subjects achieving target SBP reduction at 1 month follow up
- At 3 Months Follow Up: Percentage of subjects achieving target SBP reduction at 3 months follow up
- At 6 Months Follow Up: Percentage of subjects achieving target SBP reduction at 6 months follow up
- At 12 Month Follow Up: Percentage of subjects achieving target SBP reduction at 12 months follow up
Arm/Group | At 1 Month Follow up | At 3 Months Follow Up | At 6 Months Follow Up | At 12 Month Follow Up
Number analyzed (Participants) | 14 | 14 | 14 | 13
percentage of participants | 71.4 | 50 | 50 | 53.8

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Renal Artery Sympathetic Denervation
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Artery Sympathetic Denervation (N=19)
Arterial spasm (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2)
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.